CLINICAL TRIAL: NCT05402683
Title: Ultrasound Versus Clinical Tests as Predictors of Difficult Endotracheal Intubation in Patients With Obstructive Sleep Apnoea Undergoing Elective Surgery Under General Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amer Bahir Soliman, Amer Soliman, Tanta University
Other Study IDs: 35152/12/21
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Difficult Intubation in Obstructive Sleep Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnoea (OSA) is the most serious kind of the sleep-disordered breathing group, characterised by recurrent episodes of partial to complete obstruction of the upper airway resulting in inefficient alveolar gas exchange and desaturation[1].

It is a commonly encountered condition with a reported prevalence of 9-25% in the general population [2].

However, the majority of OSA patients presenting for surgery remain undiagnosed or untreated[3], contributing to a high rate of unexpected adverse airway outcome[4].

The various airway abnormalities represented by OSA include a large tongue, collapsible airway and crowding of the oropharyngeal structures, among others[5].

Accurate airway assessment should always be performed so as to provide appropriate planning and management of expected difficult intubation, but the common clinical screening tests (Mallampati score, inter-incisor distance, mento-hyoid distance, BMI, etc ) have shown low sensitivity and specificity with a limited predictive value, especially if only a single assessment method is used[6].

Ultrasonography could be a highly sensitive and specific tool for prediction of difficult intubation in OSA patients presented for elective surgery by measuring tongue base thickness, distance between lingual arteries, hyo-mental distance and condylar mobility.

ELIGIBILITY:
Inclusion Criteria:

1. 21-60 years old
2. ASA I, II, or III
3. STOP-BANG scoring >3

Exclusion Criteria:

* 1) Age <21 years old 2) patients with cervical spine injury, limited neck mobility, neck swelling 3) patients with lost incisor teeth 4) asymmetric mobility of the temporomandibular joint as in maxillofacial injuries/malignancies prior to surgery on the airway 5) pregnancy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be carried out on OSA patients prepared for elective surgery under general anaesthesia with tracheal intubation from Tanta University Hospitals
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound parameters | preoperative assessment
  evaluate the accuracy of the ultrasound parameters as predictors of difficult intubation in OSA patients in the perioperative period.

SECONDARY OUTCOMES:
which is better | preoperative assessment
  - To evaluate which is superior for assessment of difficult intubation in OSA patients, ultrasound or clinical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Amer AB Soliman, Bachelor, Principal Investigator — Tanta university hospitals
Locations (1):
- Tanta University hospitals, Tanta, Gharbya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided